CLINICAL TRIAL: NCT04767919
Title: Randomized Controlled Trial to Compare the Operative Outcomes and Complications of Mini-percutaneous Nephrolithotomy (Mini-PCNL) Versus Standard PCNL
Brief Title: MIP Versus PCNL for Kidney Stone Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Seth Bechis, Associate Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 191269
Record Dates: First submitted 2021-01-20; First posted 2021-02-23 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Kidney Stone
Keywords: Nephrolithotomy Laser Percutaneous Kidney Stone
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Intervention Model Description: Subjects will be assigned to one of two Standard of Care treatments for kidney stone disease and complete their treatment using one treatment modality.
Who Masked: Participant
Masking Description: Subjects will be blinded to the Standard of Care treatment they receive for their kidney stone disease
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Percutaneous Nephrolithotomy (sPCNL) (Active Comparator): The first arm will consist of a Standard of Care standard percutaneous nephrolithotomy (sPCNL)- performed using a 30 Fr access sheath following balloon dilation.
  Interventions: Procedure: Standard Percutaneous Nephrolithotomy (sPCNL)
- Minimally Invasive Percutaneous Nephrolithotomy (MIP) (Active Comparator): The second arm will consist of a Standard of Care mini percutaneous nephrolithotomy (mPCNL)- performed using an 18 Fr access sheath following either balloon dilation or dilation using a single step metal dilator.
  Interventions: Procedure: Minimally Invasive Percutaneous Nephrolithotomy (MIP)

INTERVENTIONS:
Procedure: Standard Percutaneous Nephrolithotomy (sPCNL) — Endoscopic stone procedure using a laser placed in the kidney through an 30 Fr access sheath following balloon dilation.
  Arms: Standard Percutaneous Nephrolithotomy (sPCNL)
Procedure: Minimally Invasive Percutaneous Nephrolithotomy (MIP) — Endoscopic stone procedure using a laser placed in the kidney through an 18 Fr access sheath following either balloon dilation or dilation using a single step metal dilator.
  Arms: Minimally Invasive Percutaneous Nephrolithotomy (MIP)

SUMMARY:
The decision to use standard percutaneous nephrolithotomy (PCNL) versus mini-percutaneous nephrolithotomy (MIP) has been a subject of much debate in the urological community. The investigators propose a randomized controlled trial to compare the operative outcomes and complications of mini-percutaneous nephrolithotomy (mini-PCNL) versus standard PCNL for renal stones. The results of this study will help guide the decision making regarding these two procedures in the US population and provide further insight into the utility and safety of these procedures. A cost analysis will be performed, and it is hypothesized that the reusable components of the Storz MIP set will result in lower costs of the mini-PCNL procedure compared to standard PCNL.

DETAILED DESCRIPTION:
Presurgical management will follow the standard of care and patients with active urinary tract infections will be treated prior to kidney stone surgery. After the informed consent process, the subject will be asked to complete the Wisconsin Stone Quality of Life Index (WISQOL), an externally validated and internally consistent questionnaire designed specifically for kidney stones patients. All patients should receive a computerized tomography (CT) scan prior to their procedure as standard of care for assessment of stone burden and access planning. This preoperative imaging will be assessed and scored using the standardized STONE scoring system, which has been validated for predicting treatment success and perioperative complications following PCNL.

Prior to their procedure patients will be randomized to receive one of the two interventions outlined above, only study subjects will be blinded to the randomization. Randomization will be conducted centrally for each site to ensure balance of PCNL and mini-PCNL using the CCF-Redcap randomization module to ensure proper randomization between sites. Randomization can occur at any time after enrollment prior to surgery. Study subjects will be selected from a patient pool where PCNL or mini-PCNL would be considered equally viable alternative Standard of Care procedures for treatment of kidney stone disease, with neither procedure presenting any benefit over the other. The randomization of procedure for this pool of study subjects was to guarantee that an equal number of both procedures were performed in the trial throughout all centers.

Patients choosing to participate in this research study will not be informed of which procedure they received to minimize any bias regarding postoperative pain and quality of life scores. No changes to the disclosure process will be made for any other variations or complications during their procedure outside of the research study interventions. Due to the time between the initial surgical procedure and postoperative follow-up visit there is a risk of unintentional unblinding by other providers involved with the care of study patients and access to their medical records. As such patients will be asked at the time of their follow-up visit if they remained blinded to their procedure type. Whenever possible patients should remain blinded but unblinding is not an exclusion criterion as the primary endpoint, change in hemoglobin, should not be affected by this knowledge.

A pre-operative complete blood count and basic metabolic panel will be obtained. Two endoscopic stone procedure types will be investigated in this study. The first, a standard percutaneous nephrolithotomy (sPCNL)- performed using a 30 Fr access sheath following balloon dilation. The second, a mini percutaneous nephrolithotomy (mPCNL)- performed using an 18 Fr access sheath following either balloon dilation or dilation using a single step metal dilator. Both procedures will be performed under general anesthesia with the patient in prone position. Access technique (triangulation method, ultrasound guided, or endoscopically guided) will be at the discretion of the attending surgeon. Stone lithotripter type (pneumatic, ultrasonic, or laser) and retrieval method (basket, forceps) will similarly be at the discretion of the urologist. Placement of ureteral stents will be left up to the discretion of the surgeon. Placement of nephrostomy tubes will be recorded as a protocol deviation and the indication for placement recorded. Whenever possible a single access tract will be used for the procedure and if multiple access sites are required it will be recorded as a protocol deviation. Following completion of the procedure and closure of the access tract, pressure will be applied to the surgical site for one minute. Patients with plans for a staged bilateral PCNL should only be enrolled for their first operation and should complete the quality-of-life questionnaire and imaging requirements described below prior to their second procedure.

Renal pelvis pressure monitoring is not part of the standard of care and is included as an outcome for research purposes only. There is no additional risk to the patient when monitoring this pressure and patients will be informed of this during the informed consent process.

Using a flexible cystoscope, a 5 Fr open-ended ureteral catheter will be positioned in the ureteropelvic junction for recording renal pelvis pressures. Following placement, the catheter will be secured and attached to arterial line pressure transducer positioned at the level of the kidney and connected to an invasive blood pressure (IBP) port. The arterial line pressure transducer will be fixed to IV pole at the level of the kidney and adjusted during the case if the patient bed is repositioned during the case. Transducer tubing should be flushed with normal saline to remove any air and pressure should be zeroed without any pressure being applied to the surgical site. Pressure monitoring and zeroing should be established after obtaining access but prior to active stone fragmentation or extraction and continue until closure of the access tract.

Continuous data monitoring and recording will be achieved via attaching the IBP port either on a portable vital signs monitor or the main anesthesia monitoring system. Data points should be recorded continuously whenever possible. Data will be either extracted manually from the portable monitor or automatically through the anesthesia monitoring system. Analysis of these data points to determine the mean RPP, time above >30mmHg, and maximum RPP can be conducted at the individual sites and included as part of their data set transfer or deidentified data sets can be sent to CCF for analysis of those endpoints.

Post-operatively, patients will be admitted to the hospital and monitored per usual clinical procedure. A complete blood count will be obtained on postoperative day 0, preferably in recovery, and on postoperative day 1. A basic metabolic panel will also be obtained prior to discharge. Further laboratory tests will be dictated by the patients' clinical status and length of stay. If patient length of stay exceeds one day the final complete blood count prior to discharge will also be recorded.

Along with their standard postoperative day 1 labs, an additional red topped tube (4-10ml) for IL-6 and procalcitonin will also be collected. This sample will need to be processed with several hours of collection using a centrifuge and the serum aliquots placed in cryovials prior to freezing. Individual research sites will be responsible for the lab draw, centrifuge process, freezing, and shipping of IL-6 and procalcitonin serum samples. These may be stored on site and shipped in bulk periodically or upon conclusion of patient enrollment per the preference of the study coordinator at each site. All these samples will be analyzed in bulk at the conclusion of the recruitment period.

Since higher irrigating pressures during PCNL have been linked to higher rates of the systemic inflammatory response (SIRS) this will also be included as a secondary endpoint. The criteria for SIRS will be defined as any two of the following conditions: heart rate >90 beats per minute, respiratory rate >20 respirations per minute, serum white blood cell count greater than 12,000/high power field or less than 4,000/high power field and temperature >38.0 ⁰C or <36.0 ⁰C.

Postoperative complications will be classified using the Clavien-Dindo system which has been modified for use following percutaneous nephrolithotomy. Standard of care procedures will be followed for patients requiring postoperative blood transfusions. Postoperative pain management will be left up to the discretion of the attending surgeon. The patient will be discharged from the hospital per the usual clinical protocols with a planned clinic visit between 4 and 6 weeks after surgery. In the interval following surgery readmissions, ED visits, and reoperations for study patients should be recorded.

As part of the standard of care for PCNL patients, both a renal ultrasound and a kidney, ureter, and bladder x-ray study obtained between 4 and 6 weeks postoperatively. Imaging will be reviewed by a blinded radiologist for assessment of stone free rate, defined as no visible stone fragments on either imaging set. Any discrepancies between ultrasound and x-ray modalities will be resolved with a follow-up CT scan.

If a patient receives a postoperative CT scan for another indication, this scan will take the place of the KUB and U/S for determining stone free rate. Additional data points such as parenchymal thickness at target calyx will for also be assessed for swelling/fluid accumulation.

The WISQL questionnaire, the same administered following initial consent, will be given at the 4-6 week follow-up visit to track any differences in quality of life between the two procedures. The WISQOL questionnaire specifically asks for the patients to provide answer statements that reflect their quality of life over the past four weeks. For the purposes of the second instance of the questionnaire, study subjects will be instructed to answer with respect to their symptoms since their procedure, to encompass patients who may have their follow-up visit scheduled more than four weeks from their procedure date.

The timeline for study subject participation and the required tests is presented below.

Procedures Preoperative POD0 POD1 Weeks 4-6 Informed consent X CT Scan X WISQOL Survey X X CBC X X X BMP or CMP X X Randomization X Intraoperative RPP X Serum sample (IL-6 and PCT) X KUB and renal U/S X

ELIGIBILITY:
Inclusion Criteria:

* Patients with planned PCNL and a preoperative CT scan
* Urologist obtained access and prone positioning during surgery
* Tract dilation performed either using balloon dilator or a single step mini-PCNL dilation
* Age: ≥18 years' old
* Stone size: 10-25mm
* Gender: Male and female patients
* Patients of all ethnic backgrounds
* Capable of giving informed consent
* Capable and willing to fulfill the requirements of the study
* Pre-existing indwelling nephrostomy tube or ureteral stent permitted

Exclusion Criteria:

* Anticoagulated or history of coagulopathy (with the exception of daily 81 mg aspirin)
* Conversion to open procedure
* Multiple access tracts
* Inability to give informed consent or unable to meet requirements of the study for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-06-07 (Actual); Study Completion 2024-06-07 (Actual)

PRIMARY OUTCOMES:
Blood Loss | Intraoperative period, up to 4 hours on average.
  Blood loss during study operative procedure, up to 4 hours on average, as estimated by hemoglobin levels measured immediately after surgery.

SECONDARY OUTCOMES:
Intraoperative Complication Rates | Intraoperative period, up to 4 hours on average.
  Complication rates occurring during the study operative procedure, up to 4 hours on average, including infundibular and pelvic wall tears and sheath slippage out of parenchyma, measured for all study subjects through study completion, an average of 1 year.
Renal Pressure | Intraoperative period, up to 4 hours on average.
  Operative renal pelvis pressure, measured in mm Hg, measured by a catheter placed transurethral in the ureteropelvic junction during study operative procedure, up to 4 hours on average, measured for every study subject through study completion, up to 1 year on average.
Operation Time | Intraoperative period, up to 4 hours on average.
  Length of time of study operative procedure, up to 4 hours on average, measured in hours, measured for every study subject through study completion, up to 1 year on average.
Anesthesia Time | Intraoperative period, up to 4 hours on average.
  Length of time of administration of anesthesia measured in hours during study operative procedure, up to 4 hours on average, measured for every study subject through study completion, up to 1 year on average.
Hospital Stay Time | Postoperative period, 24 hours on average.
  Length of time of stay in hospital measured in hours, beginning from time study subject leaves operating room after completion of study procedure to the time study subject is discharged from the hospital for study procedure, 24 hours on average, measured for every study subject through study completion, an average of 1 year.
Pain Medication Dose | Postoperative period, 24 hours on average.
  Dose of pain medication administered to study subject beginning from the time study subject leaves the operating room after completion of study procedure, to the time study subject is discharged from the hospital for study procedure, 24 hours on average, measured for every study subject through study completion, an average of 1 year.
Urine Output | Postoperative period, 24 hours on average.
  Volume of urine produced by study subject, measured in milliliters, beginning from time study subject leaves operating room after completion of study procedure to discharge from the hospital for study procedure, 24 hours on average, measured for every study subject through study completion, an average of 1 year.
ED Visits | Postoperative period, up to 6 weeks.
  Frequency of visits to emergency room, beginning from time study subject leaves operating room after completion of study procedure to the time study subject exits the study, up to 6 weeks, measured for every study subject through study completion, an average of 1 year.
Readmission | Postoperative period, up to 6 weeks.
  Frequency of readmission to hospital, beginning from time study subject leaves operating room after completion of study procedure to the time study subject exits the study, up to 6 weeks, measured for every study subject through study completion, an average of 1 year.
Reoperation | Postoperative period, up to 6 weeks.
  Frequency of reoperation on same side kidney as original study procedure, beginning from time study subject leaves operating room after completion of study procedure to the time study subject exits the study, up to 6 weeks, measured for every study subject through study completion, an average of 1 year.
Imaging | Postoperative period, up to 6 weeks
  Presence of stone fragments as viewed on imaging of kidney by CT scan, KUB, or ultrasound, beginning from time study subject leaves operating room after completion of study procedure to the time study subject exits the study, up to 6 weeks, measured for every study subject through study completion, an average of 1 year.
Quality of Life Questionnnaire | Postoperative period, up to 6 weeks.
  Results of Wisconsin Quality of Life Survey, measured from 1 to 5 with 1 being very true and always and 5 being not at all true and never, administered beginning from time study subject leaves operating room after completion of study procedure to the time study subject exits the study, up to 6 weeks, measured for every study subject through study completion, an average of 1 year.
IL-6 Results | Postoperative period, up to 8 hours on average.
  Measurement of Interlukin-6 in picograms per milliliters immediately after completion of study operative procedure, 0-8 hours on average, measured for every study subject through study completion, an average of 1 year.
PCT Results | Postoperative period, up to 8 hours on average.
  Measurement of procalcitonin in nanograms per milliliters immediately after completion of study procedure, 0-8 hours on average, measured for every study subject through study completion, an average of 1 year.
Pain Intensity | Postoperative period, up to 6 weeks.
  Pain measured using Stanford Pain Scale, a 0-10 scale with 10 being the greatest pain, beginning from time study subject leaves operating room after completion of study operative procedure to the time study subject exits the study, up to 6 weeks, measured for every study subject through study completion, an average of 1 year.
Postoperative Complication Rates | Postoperative period, up to 6 weeks.
  Complications rates beginning from time study subject leaves operating room after completion of study procedures to exit from study, up to 6 weeks, including fever, SIRS, blood transfusion, pleural effusions, urine leak, urinary retention, perirenal hematoma or urinoma, post-operative stent placement, ICU admission, and Clavien-Dindo Classification, measured for every study subject through study completion, an average of 1 year.
  ed study procedures
Pain Medication Frequency | [Time Frame: Postoperative period, 24 hours on average.]
  Frequency of pain medication administered to study subject beginning from the time study subject leaves the operating room after completion of study procedure, to the time study subject is discharged from the hospital for study procedure, 24 hours on average, measured for every study subject through study completion, an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Manoj Monga, M.D., Study Chair — UCSD Medical Center, San Diego
Locations (6):
- United States (5):
  - Mayo Clinic, Phoenix, Arizona
  - University of California, San Diego, Medical Center, San Diego, California
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State Unversity, Columbus, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
- University Of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Assimos D, Krambeck A, Miller NL, Monga M, Murad MH, Nelson CP, Pace KT, Pais VM Jr, Pearle MS, Preminger GM, Razvi H, Shah O, Matlaga BR. Surgical Management of Stones: American Urological Association/Endourological Society Guideline, PART I. J Urol. 2016 Oct;196(4):1153-60. doi: 10.1016/j.juro.2016.05.090. Epub 2016 May 27. PMID 27238616
- [Background] Desai MR, Sharma R, Mishra S, Sabnis RB, Stief C, Bader M. Single-step percutaneous nephrolithotomy (microperc): the initial clinical report. J Urol. 2011 Jul;186(1):140-5. doi: 10.1016/j.juro.2011.03.029. Epub 2011 May 14. PMID 21575966
- [Background] Zeng G, Wan S, Zhao Z, Zhu J, Tuerxun A, Song C, Zhong L, Liu M, Xu K, Li H, Jiang Z, Khadgi S, Pal SK, Liu J, Zhang G, Liu Y, Wu W, Chen W, Sarica K. Super-mini percutaneous nephrolithotomy (SMP): a new concept in technique and instrumentation. BJU Int. 2016 Apr;117(4):655-61. doi: 10.1111/bju.13242. Epub 2015 Aug 22. PMID 26220396
- [Background] Desai J, Solanki R. Ultra-mini percutaneous nephrolithotomy (UMP): one more armamentarium. BJU Int. 2013 Nov;112(7):1046-9. doi: 10.1111/bju.12193. Epub 2013 Jul 11. PMID 23841665
- [Background] Jackman SV, Docimo SG, Cadeddu JA, Bishoff JT, Kavoussi LR, Jarrett TW. The "mini-perc" technique: a less invasive alternative to percutaneous nephrolithotomy. World J Urol. 1998;16(6):371-4. doi: 10.1007/s003450050083. PMID 9870281
- [Background] Giusti G, Piccinelli A, Taverna G, Benetti A, Pasini L, Corinti M, Teppa A, Zandegiacomo de Zorzi S, Graziotti P. Miniperc? No, thank you! Eur Urol. 2007 Mar;51(3):810-4; discussion 815. doi: 10.1016/j.eururo.2006.07.047. Epub 2006 Aug 11. PMID 16938385
- [Background] Xu S, Shi H, Zhu J, Wang Y, Cao Y, Li K, Wang Y, Sun Z, Xia S. A prospective comparative study of haemodynamic, electrolyte, and metabolic changes during percutaneous nephrolithotomy and minimally invasive percutaneous nephrolithotomy. World J Urol. 2014 Oct;32(5):1275-80. doi: 10.1007/s00345-013-1204-2. Epub 2013 Nov 1. PMID 24177788
- [Background] Guler A, Erbin A, Ucpinar B, Savun M, Sarilar O, Akbulut MF. Comparison of miniaturized percutaneous nephrolithotomy and standard percutaneous nephrolithotomy for the treatment of large kidney stones: a randomized prospective study. Urolithiasis. 2019 Jun;47(3):289-295. doi: 10.1007/s00240-018-1061-y. Epub 2018 Jun 1. PMID 29858913
- [Background] Sakr A, Salem E, Kamel M, Desoky E, Ragab A, Omran M, Fawzi A, Shahin A. Minimally invasive percutaneous nephrolithotomy vs standard PCNL for management of renal stones in the flank-free modified supine position: single-center experience. Urolithiasis. 2017 Dec;45(6):585-589. doi: 10.1007/s00240-017-0966-1. Epub 2017 Feb 22. PMID 28229197
- [Background] Cheng F, Yu W, Zhang X, Yang S, Xia Y, Ruan Y. Minimally invasive tract in percutaneous nephrolithotomy for renal stones. J Endourol. 2010 Oct;24(10):1579-82. doi: 10.1089/end.2009.0581. PMID 20839954
- [Background] Zhong W, Zeng G, Wu W, Chen W, Wu K. Minimally invasive percutaneous nephrolithotomy with multiple mini tracts in a single session in treating staghorn calculi. Urol Res. 2011 Apr;39(2):117-22. doi: 10.1007/s00240-010-0308-z. Epub 2010 Sep 7. PMID 20821200
- [Background] Mishra S, Kurien A, Ganpule A, Muthu V, Sabnis R, Desai M. Percutaneous renal access training: content validation comparison between a live porcine and a virtual reality (VR) simulation model. BJU Int. 2010 Dec;106(11):1753-6. doi: 10.1111/j.1464-410X.2010.09753.x. Epub 2010 Oct 15. PMID 20950308
- [Background] Wu C, Hua LX, Zhang JZ, Zhou XR, Zhong W, Ni HD. Comparison of renal pelvic pressure and postoperative fever incidence between standard- and mini-tract percutaneous nephrolithotomy. Kaohsiung J Med Sci. 2017 Jan;33(1):36-43. doi: 10.1016/j.kjms.2016.10.012. Epub 2016 Dec 22. PMID 28088272
- [Background] Karami H, Gholamrezaie HR. Totally tubeless percutaneous nephrolithotomy in selected patients. J Endourol. 2004 Jun;18(5):475-6. doi: 10.1089/0892779041271580. PMID 15253824
- [Background] Alsyouf M, Abourbih S, West B, Hodgson H, Baldwin DD. Elevated Renal Pelvic Pressures during Percutaneous Nephrolithotomy Risk Higher Postoperative Pain and Longer Hospital Stay. J Urol. 2018 Jan;199(1):193-199. doi: 10.1016/j.juro.2017.08.039. Epub 2017 Aug 12. PMID 28807646
- [Background] Kukreja RA, Desai MR, Sabnis RB, Patel SH. Fluid absorption during percutaneous nephrolithotomy: does it matter? J Endourol. 2002 May;16(4):221-4. doi: 10.1089/089277902753752160. PMID 12042103
- [Background] Loftus CJ, Hinck B, Makovey I, Sivalingam S, Monga M. Mini Versus Standard Percutaneous Nephrolithotomy: The Impact of Sheath Size on Intrarenal Pelvic Pressure and Infectious Complications in a Porcine Model. J Endourol. 2018 Apr;32(4):350-353. doi: 10.1089/end.2017.0602. PMID 29385812
- [Background] Zhong W, Zeng G, Wu K, Li X, Chen W, Yang H. Does a smaller tract in percutaneous nephrolithotomy contribute to high renal pelvic pressure and postoperative fever? J Endourol. 2008 Sep;22(9):2147-51. doi: 10.1089/end.2008.0001. PMID 18811571
- [Background] Rettig TC, Verwijmeren L, Dijkstra IM, Boerma D, van de Garde EM, Noordzij PG. Postoperative Interleukin-6 Level and Early Detection of Complications After Elective Major Abdominal Surgery. Ann Surg. 2016 Jun;263(6):1207-12. doi: 10.1097/SLA.0000000000001342. PMID 26135695
- [Background] Omar M, Noble M, Sivalingam S, El Mahdy A, Gamal A, Farag M, Monga M. Systemic Inflammatory Response Syndrome after Percutaneous Nephrolithotomy: A Randomized Single-Blind Clinical Trial Evaluating the Impact of Irrigation Pressure. J Urol. 2016 Jul;196(1):109-14. doi: 10.1016/j.juro.2016.01.104. Epub 2016 Feb 8. PMID 26869311
- [Background] Tefekli A, Ali Karadag M, Tepeler K, Sari E, Berberoglu Y, Baykal M, Sarilar O, Muslumanoglu AY. Classification of percutaneous nephrolithotomy complications using the modified clavien grading system: looking for a standard. Eur Urol. 2008 Jan;53(1):184-90. doi: 10.1016/j.eururo.2007.06.049. Epub 2007 Jul 24. PMID 17651892
- [Background] Okhunov Z, Friedlander JI, George AK, Duty BD, Moreira DM, Srinivasan AK, Hillelsohn J, Smith AD, Okeke Z. S.T.O.N.E. nephrolithometry: novel surgical classification system for kidney calculi. Urology. 2013 Jun;81(6):1154-9. doi: 10.1016/j.urology.2012.10.083. Epub 2013 Mar 26. PMID 23540858
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Michel MS, Trojan L, Rassweiler JJ. Complications in percutaneous nephrolithotomy. Eur Urol. 2007 Apr;51(4):899-906; discussion 906. doi: 10.1016/j.eururo.2006.10.020. Epub 2006 Oct 25. PMID 17095141
- [Background] Bucuras V, Gopalakrishnam G, Wolf JS Jr, Sun Y, Bianchi G, Erdogru T, de la Rosette J; CROES PCNL Study Group. The Clinical Research Office of the Endourological Society Percutaneous Nephrolithotomy Global Study: nephrolithotomy in 189 patients with solitary kidneys. J Endourol. 2012 Apr;26(4):336-41. doi: 10.1089/end.2011.0169. Epub 2011 Oct 17. PMID 22004844